CLINICAL TRIAL: NCT05127434
Title: A Phase 2/3, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus (RSV), in Adults ≥60 Years of Age
Brief Title: A Study to Evaluate the Safety and Efficacy of mRNA-1345 Vaccine Targeting Respiratory Syncytial Virus (RSV) in Adults ≥60 Years of Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P301; 2021-005026-20 (EudraCT Number)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Respiratory syncytial virus; Safety; Vaccines
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- mRNA-1345 (Experimental): Single injection of mRNA-1345 on Day 1.
  Interventions: Drug: mRNA-1345
- Placebo (Experimental): Single injection of mRNA-1345 matching-placebo on Day 1.
  Interventions: Drug: Placebo
- mRNA-1345 BD (Experimental): Single injection of mRNA-1345 on BD Day 1.
  Interventions: Drug: mRNA-1345

INTERVENTIONS:
Drug: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo
Drug: mRNA-1345 — Sterile liquid for injection
  Arms: mRNA-1345; mRNA-1345 BD

SUMMARY:
The main purpose of Part A of this study is to evaluate the safety and tolerability of mRNA-1345 vaccine and to demonstrate the efficacy of a single dose of mRNA-1345 vaccine in the prevention of a first episode of RSV-associated lower respiratory tract disease (RSV-LRTD) as compared with placebo from 14 days postinjection through 12 months.

The main purpose of Part B of this study is to evaluate the safety, tolerability and immunogenicity of a booster dose (BD) of mRNA-1345 administered 24 months after the primary dose.

DETAILED DESCRIPTION:
The study will be conducted in 2 phases: Phase 2 and Phase 3. In the Part A Phase 2 segment, up to 2,000 participants will be randomly assigned to receive a single injection of either mRNA-1345 vaccine at the selected dose or placebo in a 1:1 randomization ratio.

In the Part A Phase 3 segment, approximately 35,000 participants will be randomly assigned to receive a single injection of either mRNA-1345 vaccine at the selected dose or placebo in a 1:1 randomization ratio.

In the Part B substudy, 1500 participants who received a dose of mRNA-1345 in Part A Phase 3 will be randomly assigned in a 2:1 randomization ratio to receive a single BD injection of either mRNA-1345 at the selected dose or placebo.

ELIGIBILITY:
Key Inclusion Criteria (Part A):

* Adults ≥ 60 years of age who are primarily responsible for self-care and activities of daily living. Participants may have one or more chronic medical diagnoses (including chronic heart failure [CHF] and chronic obstructive pulmonary disease [COPD]), but should be medically stable
* Body mass index from ≥18 kilograms (kg)/square meter (m^2) to ≤35 kg/m^2

Key Inclusion Criteria (Part B):

* Randomized to and were subsequently vaccinated with the mRNA-1345 study injection in Part A at least 21 months prior to Screening.

Key Exclusion Criteria (Part A):

* Participation in another clinical research study where participant has received an investigational product (drug/biologic/device) within 6 months before the planned date of the Day 1 study injection.
* Current participation in research involving receipt of any investigational RSV product
* History of a serious reaction to any prior vaccination or Guillain-Barré syndrome within 6 weeks of any prior influenza immunization.
* Received or plans to receive any non-study vaccine within 28 days before or after the Day 1 study injection.

Key Exclusion Criteria (Part B):

* Participation in another clinical research study where participant has received an investigational product (drug/biologic/device) within 6 months before the planned date of BD study injection (BD Day 1).
* History of a serious reaction to any prior vaccination, or Guillain-Barré syndrome within 6 weeks of any prior influenza immunization.
* Received or plans to receive any non-study vaccine (including authorized or approved vaccines for the prevention of coronavirus disease 2019 (COVID-19) regardless of type of vaccine) within 14 days before or after the BD Day 1 study injection.
* Received or plans to receive any commercial RSV vaccination at any time prior to BD study injection (BD Day 1) or during the substudy.

Other inclusion and/or exclusion criteria may apply.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36814 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to 7 days after each injection
Number of Participants with Unsolicited Adverse Events (AEs) | Up to 28 days after each injection
Number of Participants With Medically Attended AEs (MAAEs), Adverse Events of Special Interests (AESIs), Serious Adverse Events (SAEs), and AEs Leading to Withdrawal | Up to BD Day 181
Vaccine Efficacy (VE) of mRNA-1345 to Prevent a First Episode of RSV-LRTD with 2 or More Symptoms | From 14 days postinjection up to 12 months postinjection
  VE of mRNA-1345 to prevent reverse transcription polymerase chain reaction (RT-PCR) confirmed protocol-defined RSV-LRTD, defined as 100*(1-HR ratio), where HR is the hazard ratio (mRNA-1345 versus placebo).
VE of mRNA-1345 to Prevent a First Episode of RSV-LRTD with 3 or More Symptoms | From 14 days postinjection up to 12 months postinjection
  VE of mRNA-1345 to prevent reverse transcription polymerase chain reaction (RT-PCR) confirmed protocol-defined RSV-LRTD, defined as 100*(1-HR ratio), where HR is the hazard ratio (mRNA-1345 versus placebo).
Geometric Mean Titer (GMT) of Serum Respiratory Syncytial Virus Subtype A (RSV-A) and Respiratory Syncytial Virus Subtype B (RSV-B) Neutralizing Antibodies | BD Day 29
Geometric Mean Ratio (GMR) of Serum RSV-A and RSV-B Neutralizing Antibodies After BD Compared to After Initial Dose | BD Day 29

SECONDARY OUTCOMES:
VE of mRNA-1345 to Prevent a First Episode of RSV-Associated Acute Respiratory Disease (RSV-ARD) | From 14 days postinjection up to 12 months postinjection
  VE of mRNA-1345 to prevent RT-PCR confirmed protocol-defined RSV-ARD, defined as 100*(1-HR ratio), where HR is the hazard ratio (mRNA-1345 versus placebo).
VE of mRNA-1345 to Prevent First Hospitalization Associated with RSV-ARD or RSV-LRTD | From 14 days postinjection up to 12 months postinjection
  VE of mRNA-1345 to prevent first hospitalization associated with RSV-ARD or RSV-LRTD, defined as 100*(1-HR ratio), where HR is the hazard ratio (mRNA-1345 versus placebo).
GMT of Serum RSV Neutralizing Antibodies | Baseline through up to 24 months postinjection
Geometric Mean Concentration (GMC) of Serum RSV Binding Antibodies | Baseline through up to 24 months postinjection
Seroresponse Rate in RSV Neutralizing Antibodies | Baseline through up to 24 months postinjection
Geometric Mean Fold-Rise (GMFR) of Postbaseline/Baseline Antibody Titers | Baseline through up to 24 months postinjection
Proportion of Participants with ≥4-fold Increases in Antibody Titers from Baseline | Baseline through up to 24 months postinjection
Seroresponse Rate (SRR) Difference Between Serum RSV-A and RSV-B Neutralizing Antibodies After BD Compared to After Initial Dose | BD Day 29
GMT of Serum RSV-A and RSV-B Neutralizing Antibodies | BD Day 1 and Day 181
GMFR of Serum RSV-A and RSV-B Neutralizing Antibodies from Pre-primary Dose (Baseline) | Baseline, BD Day 1, Day 29 and Day 181
SRR of Serum RSV-A and RSV-B Neutralizing Antibodies from Pre-primary Dose (Baseline) | Baseline, BD Day 1, Day 29 and Day 181

CONTACTS AND LOCATIONS:
Locations (268):
- United States (132):
  - AES - DRS - Synexus Clinical Research US, Inc. - Birmingham, Birmingham, Alabama
  - Accel Research Site - Achieve - Birmingham, Birmingham, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - AES - DRS - Optimal Research Alabama - Huntsville, Huntsville, Alabama
  - Hope Research Institute LLC - Hunt - PPDS, Hunt, Arizona
  - Desert Clinical Research, LLC - CCT, Mesa, Arizona
  - Hope Research Institute LLC - Phoenix - Hunt - PPDS, Phoenix, Arizona
  - AES - DRS - Synexus Clinical Research US, Inc. - Phoenix Central, Phoenix, Arizona
  - Synexus Clinical Research US, Inc. - Phoenix Southeast, Phoenix, Arizona
  - Tucson Neuroscience Research - M3 WR, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Velocity Clinical Research, Banning, Banning, California
  - Hope Clinical Research, LLC, Canoga Park, California
  - Velocity Clinical Research - Chula Vista - PPDS, Chula Vista, California
  - PPD Virtual - Science 37, Inc, Culver City, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - PRI, LLC - Los Alamitos - M3 WR, Los Alamitos, California
  - PRI, LLC - Newport Beach - M3 WR, Newport Beach, California
  - FOMAT Medical Research - FOMAT - HyperCore - PPDS, Oxnard, California
  - Reddy Care Medical, Pomona, California
  - Paradigm Clinical Research Institute Inc - ClinEdge - PPDS, Redding, California
  - Medical Center For Clinical Research - M3 WR, San Diego, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Tekton Research - Fort Collins - PPDS, Fort Collins, Colorado
  - Tekton Research - Longmont - PPDS, Longmont, Colorado
  - Paradigm Clinical Research Institute Inc - ClinEdge - PPDS, Wheat Ridge, Colorado
  - Clinical Research Consultants LLC - ClinEdge - PPDS, Milford, Connecticut
  - Washington Health Institute, Washington D.C., District of Columbia
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Fleming Island Clinical Research Center, Fleming Island, Florida
  - Velocity Clinical Research - Hallandale Beach - PPDS, Hallandale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc. M3 WR, Lake City, Florida
  - Accel Research Sites - Maitland - ERN - PPDS, Maitland, Florida
  - Spotlight Research Center, LLC, Miami, Florida
  - IMA Clinical Research - Manhattan - PPDS, Miami Beach, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - The Villages, Orlando, Florida
  - Health Awareness Inc, Port Saint Lucie, Florida
  - IMA Clinical Research - Saint Petersburg - PPDS, St. Petersburg, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Petersburg, St. Petersburg, Florida
  - Clinical Trials of Tampa, Tampa, Florida
  - Palm Beach Research - ClinEdge - PPDS, West Palm Beach, Florida
  - Clinical Site Partners - Winter Park - HyperCore -PPDS, Winter Park, Florida
  - Mount Vernon Clinical Research, LLC - M3 WR, Atlanta, Georgia
  - Masters of Clinical Research Inc, Augusta, Georgia
  - Centricity Research - Roswell - HyperCore - PPDS, Columbus, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Javara, Inc./Privia Medical Group Georgia, LLC, Fayetteville, Georgia
  - Drug Studies America - ClinEdge - PPDS, Marietta, Georgia
  - Randomize Now -Commerce Dr, Peachtree City, Georgia
  - Velocity Clinical Research (Savannah - Georgia) - PPDS, Savannah, Georgia
  - Clinical Research Atlanta - ERN-PPDS, Stockbridge, Georgia
  - East West Medical Research Institute, Honolulu, Hawaii
  - Velocity Clinical Research - Boise - PPDS, Meridian, Idaho
  - AES - DRS - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - Affinity Health (Oak Brook), Oak Brook, Illinois
  - DM Clinical - Chicago, River Forest, Illinois
  - AES - DRS - Synexus Clinical Research US, Inc. - Evansville, Evansville, Indiana
  - Velocity Clinical Research - Valparaiso - PPDS, Valparaiso, Indiana
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Versailles Family Medicine - CCT - PPDS, Versailles, Kentucky
  - Velocity Clinical Research (Baton Rouge - Louisiana) - PPDS, Baton Rouge, Louisiana
  - Benchmark Research - Covington - HyperCore - PPDS, Covington, Louisiana
  - Benchmark Research - Metairie - HyperCore - PPDS, Metairie, Louisiana
  - IMA Clinical Research - Monroe, LA - PPDS, Monroe, Louisiana
  - DelRicht Clinical Research, LLC - Internal - Covington - PPDS, New Orleans, Louisiana
  - Privia Medical Group, LLC - Annapolis - Javara - PPDS, Annapolis, Maryland
  - CBH Health - CenExel CBH - PPDS, Gaithersburg, Maryland
  - Velocity Clinical Research (Rockville - Maryland) - PPDS, Rockville, Maryland
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research - Southfield - ERN - PPDS, Southfield, Michigan
  - Clinical Research Institute, Inc - CRN - PPDS, Minneapolis, Minnesota
  - AES - DRS - Synexus Clinical Research US, Inc. - Minneapolis, Richfield, Minnesota
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Louis, Creve Coeur, Missouri
  - Montana Medical Research, Missoula, Montana
  - Boeson Research MSO - Missoula - ERN - PPDS, Missoula, Montana
  - Skyline Medical Center, PC - CCT Research, Elkhorn, Nebraska
  - Methodist Physicians Clinic - CCT Research - PPDS, Fremont, Nebraska
  - Velocity Clinical Research (Grand Island - Nebraska) - PPDS, Grand Island, Nebraska
  - Velocity Clinical Research (Lincoln - Nebraska) - PPDS, Lincoln, Nebraska
  - Velocity Clinical Research (Omaha - Nebraska) - PPDS, Omaha, Nebraska
  - CCT Research, Papillion, Nebraska
  - HEALOR Primary Care - Physicians Las Vegas - CCT, Las Vegas, Nevada
  - Excel Clinical Research - Las Vegas, Las Vegas, Nevada
  - IMA Clinical Research - Raritan - PPDS, Raritan, New Jersey
  - Riverside Medical Group - Circuit - PPDS, Secaucus, New Jersey
  - Velocity Clinical Research - East Syracuse - PPDS, East Syracuse, New York
  - Velocity Clinical Research (Endwell - New York) - PPDS, Endwell, New York
  - Drug Trials America, Hartsdale, New York
  - AES - DRS - Synexus Clinical Research US, Inc. - New York, New York, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Carolina Institute for Clinical Research - M3 WR, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - CTI Clinical Research, Cincinnati, Ohio
  - Velocity Clinical Research (Cincinnati - Ohio) - PPDS, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati - PPDS, Cincinnati, Ohio
  - AES - DRS - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - Tekton Research - Oklahoma - PPDS, Edmond, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Summit Research Network, Inc. - Portland - Headlands - PPDS, Portland, Oregon
  - Hatboro Medical Associates - CCT - PPDS, Hatboro, Pennsylvania
  - DM Clinical Research - Philadelphia - ERN - PPDS, Philadelphia, Pennsylvania
  - Velocity Clinical Research (Dakota Dunes - South Dakota) - PPDS, Dakota Dunes, South Dakota
  - American Indian Clinical Trials Research Network, Rapid City, South Dakota
  - Affinity Health - Nashville, Nashville, Tennessee
  - Premier Family Physicians - Austin - Hunt - PPDS, Austin, Texas
  - Tekton Research, Austin, Texas
  - PanAmerican Clinical Research LLC, Brownsville, Texas
  - ACRC Trials - Carrollton - Hunt - PPDS, Carrollton, Texas
  - Privia Medical Group- North Texas - West Parker Road - Fort Worth - Javara - PPDS, Fort Worth, Texas
  - Allure Health LLC, Friendswood, Texas
  - Olympus Family Medicine- CCT, Friendswood, Texas
  - Village Health Partners Frisco Medical Village, Frisco, Texas
  - West Houston Clinical Research - Hunt - PPDS, Houston, Texas
  - DM Clinical Research - Bellaire - ERN - PPDS, Houston, Texas
  - DM Clinical-TCDD, Humble, Texas
  - Helios CR, Inc. - Houston - PPDS, Keller, Texas
  - AIM Trials, Plano, Texas
  - AES - DRS - Synexus Clinical Research US, Inc. - San Antonio, San Antonio, Texas
  - Clinical Trials of Texas, LLC - HyperCore - PPDS, San Antonio, Texas
  - Privia Medical Group- North Texas - Stephenville - Javara - PPDS, Stephenville, Texas
  - DM Clinical Research - Sugarland - ERN - PPDS, Sugar Land, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - DM Clinical Research - ERN, Tomball, Texas
  - Cope Family Medicine - CCT - PPDS, Bountiful, Utah
  - Alpine Research Organization, Inc, Clinton, Utah
  - South Ogden Family Medicine - CCT, South Ogden, Utah
  - Health Research of Hampton Roads Inc., Newport News, Virginia
  - Velocity Clinical Research - Family Practice - Portsmouth - PPDS, Portsmouth, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Seattle Clinical Research Center, Seattle, Washington
- Argentina (5):
  - Instituto Medico Platense, Buenos Aires, Provincial de Buenos Aires
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Ciudad Autónoma de BuenosAires
  - Fundación Dr. Mario Socolinsky - Centro de Vacunación Proteger, Ciudad Autónoma de BuenosAires
  - Centro Medico Barrio Parque, Ciudad Autónoma de BuenosAires
  - Consultorios Médicos Dr. Doreski, Ciudad Autónoma de BuenosAires
- Australia (6):
  - Paratus Clinical Research - Canberra - PPDS, Bruce, Australian Capital Territory
  - Paratus Clinical Research - Western Sydney - PPDS, Blacktown, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Northside Health, Coffs Harbour, New South Wales
  - Holdsworth House Medical Brisbane, Fortitude Valley, Queensland
  - Emeritus Research - PPDS, Camberwell, Victoria
- Bangladesh (4):
  - JHU-Projahnmo Zakiganj site, Zakiganj, Sylhet Division
  - icddr,b Matlab Health Research Center, Chāndpur
  - Icddr,b Kamalapur Field Site, Dhaka
  - JHU-Projahnmo Sylhet site, Sylhet
- Belgium (4):
  - ANIMA Research Center, Diepenbeek
  - Vaccinopolis, Edegem
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - Ziekenhuis Oost-Limburg, Genk
- Canada (10):
  - CARe Clinic, Red Deer, Alberta
  - Okanagan Clinical Trials - Headlands - PPDS, Kelowna, British Columbia
  - Centricity Research - Toronto - HyperCore - PPDS, Etobicoke, Ontario
  - Dr. Steven Z. Zizzo Medicine Professional Corporation, Hamilton, Ontario
  - LMC Clinical Research Inc (Bayview), Toronto, Ontario
  - Centricity Research - Quebec - HyperCore - PPDS, Lévis, Quebec
  - Diex Recherche - Joilette - PPDS, Saint-Charles-Borromée, Quebec
  - Diex Recherche - Sherbrooke - PPDS, Sherbrooke, Quebec
  - Diex Recherche - Trois Rivieres - PPDS, Trois-Rivières, Quebec
  - Diex Recherche - Québec - PPDS, Québec
- Chile (5):
  - Hospital Base de Osorno, Osorno, Los Lagos Region
  - Centro de Investigacion del Maule, Talca, Maule Region
  - Centro Respiratorio Integral LTDA. (CENRESIN), Quillota, Región de Valparaíso
  - Biomedica Research Group, Santiago, Santiago Metropolitan
  - BIOCINETIC SpA, Santiago, Santiago Metropolitan
- Colombia (10):
  - Institucion Clinica de la Costa SAS, Barranquilla, Atlántico
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Aguazul, Aguazul, Casanare Department
  - Solano & Terront Servicios Médicos LTDA (UNIENDO) Bogota, Bogota, Cundinamarca
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Bogota, Bogota, Cundinamarca
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Chia, Chía, Cundinamarca
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Girardot, Girardot City, Cundinamarca
  - IPS Centro de Investigacion Clinicas Cardiomet, Pereira, Risaralda Department
  - Fundacion Oftalmologica de Santander Foscal, Floridablanca, Santandar
  - Centro de Atención e Investigación Médica S.A. - CAIMED - Ibague, Ibagué, Tolima Department
  - Centro Medico Imbanaco de Cali S.A., Cali, Valle de Cuaca
- Costa Rica (4):
  - Campus Universidad EARTH, finca La Flor, Liberia, Guanacaste Province
  - Instituto de Investigación en Ciencias Médicas S.A., San José
  - Hospital CIMA San Jose, San José
  - Hospital Clínica Bíblica Sede Santa Ana, San José
- Finland (10):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Järvenpää Vaccine Research Clinic, Jarvenpaa
  - KokkolaVaccine Research Clinic, Kokkola
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turku Vaccine Research Clinic, Turku
- Germany (6):
  - AES - DRS - Synexus Frankfurt Research Centre, Frankfurt am Main, Hesse
  - Infektioresearch GmbH & Co. KG, Frankfurt am Main, Hesse
  - Klinische Forschung Hannover-Mitte GmbH, Hanover, Lower Saxony
  - Klinische Forschung, Schwerin GmbH (KFGN), Schwerin, Mecklenburg-West Pomerania
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - AES - DRS - Synexus Berlin Research Centre, Berlin
- Japan (10):
  - Fukui General Clinic, Fukui-shi, Fukui
  - Tenjin Sogo Clinic, Fukuoka, Fukuoka
  - Boocs Clinic Fukuoka, Hakata-ku, Fukuoka
  - Motomachi Takatsuka Naika Clinic, Naka-ku, Yokohama-ku, Kanagawa
  - Medical Corporation Asbo Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - Higashi Shinjuku Clinic, Shinjuku-ku, Tokyo
  - NewHeart Watanabe Institute, Suginami-ku, Tokyo
  - Sekino Hospital, Toshima-ku, Tokyo
  - SOUSEIKAI PS Clinic, Fukuoka
- Mexico (7):
  - AES - AS - RM Pharma Specialists Mexico City, Ciudad de Mexcio, Ciudad de Mexcio
  - AES - AS - CEMDEC Mexico City, Ciudad de Mexcio, Ciudad de Mexcio
  - Maria del rayo morfin otero, Guadalajara, Jalisco
  - Accelerium, S. de R.L. de C.V., Monterrey, Nuevo León
  - Investigacion en Salud y Metabolismo S.C., Chihuahua City
  - Hospital General 450, Durango
  - PanAmerican Clinical Research-Avenida, Querétaro
- New Zealand (6):
  - Southern Clinical Trials Limited, Christchurch, Canterbury
  - Lakeland Clinical Trials, Rotorua, Canterbury
  - Southern Clinical Trials Waitemata, Auckland
  - New Zealand Clinical Research - Auckland, Auckland
  - Optimal Clinical Trials Ltd, Auckland
  - Southern Clinical Trials - Tasman, Nelson
- Panama (2):
  - CEVAXIN Avenida México, Panama City, Calidonia
  - CEVAXIN 24 de diciembre, Panama City
- Poland (6):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Silesian Voivodeship
  - Ostrowieckie Centrum Medyczne Spólka Cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Puerto Rico (3):
  - BRCR Global Puerto Rico (Ponce), Ponce
  - Caribbean Medical Research Center, San Juan
  - Proyecto ACTU, San Juan
- Singapore General Hospital (SGH), Singapore, Singapore
- South Africa (6):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Dr. J Breedt, Pretoria, Gauteng
  - AES - DRS - Synexus - Stanza Clinical Research Centre, Pretoria, Gauteng
  - AES - DRS - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Aliwal Shoal Medical Center, eMkhomazi, KwaZulu-Natal
  - AES - DRS - Synexus - Helderberg Clinical Research Centre, Somerset West, Western Cape
- South Korea (11):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inha University Hospital, Jung-gu, Incheon
  - Samsung Medical Center - PPDS, Gangnam-gu, Seoul
  - Ewha Womans University Seoul Hospital, Gangseo-gu, Seoul
  - Dong-A University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Soon Chun Hyang University Hospital Bucheon, Gyeonggi-do
  - Catholic Kwandong University International St. Mar, Incheon
  - Severance Hospital Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (5):
  - ABS Centelles, Centelles, Barcelona
  - Hospital Son Llatzer, Son Ferriol, Palma de Mallorca
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - FISABIO Oftalmología Médica (FOM), Valencia
- Taiwan (4):
  - China Medical University Hospital - PPDS, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (11):
  - Bristol Royal Infirmary, Bristol, Avon
  - AES - DRS - NW Consortium Lancashire, Chorley, Lancashire
  - AES - DRS - Synexus Hexham Clinical Research Centre, Hexham, Northumberland
  - Cheadle Hospital, Stoke-on-Trent, Staffordshire
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - AES - DRS - Synexus Scotland Clinical Research Centre, Bellshill
  - AES - DRS - Synexus Midlands Clinical Research Centre, Birmingham
  - Layton Medical Centre, Blackpool
  - AES - DRS - Synexus Wales Clinical Research Centre, Cardiff
  - AES - DRS - NW Consortium Merseyside, Liverpool
  - AES - DRS - NW Consortium Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goswami J, Baqui AH, Doreski PA, Perez Marc G, Jimenez G, Ahmed S, Zaman K, Duncan CJA, Ujiie M, Ramet M, Perez-Breva L, Lan L, Du J, Kapoor A, Mehta S, Tomassini JE, Huang W, Zhou H, Stoszek SK, Priddy F, Lin N, Le Cam N, Shaw CA, Slobod K, Wilson E, Miller JM, Das R. Humoral Immunogenicity of mRNA-1345 RSV Vaccine in Older Adults. J Infect Dis. 2024 Nov 15;230(5):e996-e1006. doi: 10.1093/infdis/jiae316. PMID 38889247
- [Derived] Wilson E, Goswami J, Baqui AH, Doreski PA, Perez-Marc G, Zaman K, Monroy J, Duncan CJA, Ujiie M, Ramet M, Perez-Breva L, Falsey AR, Walsh EE, Dhar R, Wilson L, Du J, Ghaswalla P, Kapoor A, Lan L, Mehta S, Mithani R, Panozzo CA, Simorellis AK, Kuter BJ, Schodel F, Huang W, Reuter C, Slobod K, Stoszek SK, Shaw CA, Miller JM, Das R, Chen GL; ConquerRSV Study Group. Efficacy and Safety of an mRNA-Based RSV PreF Vaccine in Older Adults. N Engl J Med. 2023 Dec 14;389(24):2233-2244. doi: 10.1056/NEJMoa2307079. PMID 38091530